CLINICAL TRIAL: NCT03559348
Title: Phase II Trial of Biweekly S-1, Leucovorin and Gemcitabine in Elderly Patients With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); China Medical University Hospital (Other); Kaohsiung Medical University (Other); Chang Gung Memorial Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1217
Record Dates: First submitted 2018-04-18; First posted 2018-06-18 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: in Elderly Patients
MeSH Terms: interventions — Leucovorin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biweekly TS-1, Leucovorin and Gemcitabine (GSL) (Experimental): Gemcitabine 800 mg/m2 , on day 1 S-1 80, 100 or 120 mg/d, orally twice daily on day 1 to 7 Leucovorin 60 mg/d, orally twice daily on day 1 to 7 Every 14 days as one cycle
  Interventions: Drug: chemotherapy: TS-1, Leucovorin and Gemcitabine

INTERVENTIONS:
Drug: chemotherapy: TS-1, Leucovorin and Gemcitabine — Gemcitabine 800 mg/m2 , on day 1 S-1 80, 100 or 120 mg/d, orally twice daily on day 1 - 7; Leucovorin 60 mg/d, orally twice daily on day 1 - 7; Every 14 days as one cycle.

SUMMARY:
Multiple centers, uncontrolled, open-label, non-randomized single-arm study

DETAILED DESCRIPTION:
To evaluate the following items in patients with metastatic pancreatic adenocarcinoma receiving GSL treatment, Primary objective: Overall tumor response rate (by RECIST criteria)

Secondary objectives:

Disease control rate (Objective response rate + stable disease ≧ 16 weeks) Time to tumor progression Progression-free survival Overall survival Clinical benefit response Quality of life Safety profile Biomarker of pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have cyto-/histologically confirmed, recurrent or metastatic adenocarcinoma of the pancreas.
2. Patients have disease measurable or evaluable on x-ray, computed tomography scan, or physical examination.
3. Patients have no history of prior chemotherapy for metastatic pancreatic cancer. Patients who had received chemotherapy as in an adjuvant or neoadjuvant setting which was completed at least 6 months before recurrence are eligible.
4. Patients with prior radiotherapy are eligible if the irradiated area does not involve the only lesion of measurable / evaluable disease.
5. Baseline ECOG performance status is 2.
6. Patients have life expectancy of at least 12 weeks.
7. Patients have age 70 years.
8. Patients have adequate organ function.
9. Patients with biliary obstruction which is adequate drained before enrollment are eligible.
10. Patients agree to have an indwelling venous catheter implanted.
11. Women or men of reproductive potential should agree to use an effective contraceptive method.
12. All patients must be informed of the investigational nature of this study and must sign written informed consents.

Exclusion Criteria:

1. Patients who have major abdominal surgery, radiotherapy or other investigating agents within 4 weeks are not eligible. Patients who have palliative radiotherapy for bony metastasis will be eligible if the irradiated area does not involve the only lesion of measurable / evaluable disease.
2. Patients with metastatic lesion in central nervous system.
3. Patients with active infection.
4. Patients with active cardiopulmonary disease or history of ischemic heart disease.
5. Patients who have peripheral neuropathy > grade I of any etiology.
6. Patients who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, cirrhosis of the liver, and the rest will be at the discretion of in-charged investigator.
7. Patients who have other prior or concurrent malignancy except for adequately treated in situ carcinoma of cervix or adequately.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 5.0 months
  The progression-free survival time for elderly patients with advanced pancreatic cancer

SECONDARY OUTCOMES:
Overall tumor response rate | up to 18 months

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Chang-Gung Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided